CLINICAL TRIAL: NCT04407468
Title: Awake Prone Positioning and Oxygen Therapy in Patients With COVID-19 (APRONOX)
Brief Title: Awake Prone Positioning and Oxygen Therapy in Patients With COVID-19
Acronym: APRONOX
Status: Completed | Type: Observational
Sponsor: Hospital General San Juan del Rio (Network)
Collaborators: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Orlando Rubén Pérez-Nieto, Dr. Orlando Ruben Perez Nieto, Hospital General San Juan del Rio
Other Study IDs: 1178/SESEQ-HSGJR/08-05-20/UTI
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: COVID; ARDS; Pneumonia
Keywords: COVID; ARDS; PRONE POSITION
MeSH Terms: conditions — Pneumonia | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID: Patients with or without prone position
  Interventions: Procedure: Prone position

INTERVENTIONS:
Procedure: Prone position — Position of the patient in which he is face down, for an improvement in oxygenation

SUMMARY:
The prone position strategy for patients with acute respiratory distress syndrome (ARDS) is simple and cost-effective from the first description on its use in patients with acute respiratory failure to improve hypoxemia. Different studies have investigated its safety and efficacy in various clinical settings, demonstrating that its early use in combination with non-invasive mechanical ventilation (NIV) or high-flow oxygen therapy can reduce intubation rate and mortality in ARDS. In the Coronavirus disease 2019 (COVID-19) pandemic, high-value medicine and resource optimization are critical.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a pandemic that has significantly challenged health systems worldwide. Due to the large number of infections around the world, the implementation of strategies to reduce the number of intubations and the need for invasive mechanical ventilation becomes important. In addition to the inability of the Mexican health system to respond, patients under invasive ventilation have not had a favorable survival outcome. Up to 97% mortality has been reported in patients requiring intubation. The exact cause of this poor prognosis is not yet known. Early recognition of hypoxemic patients could help with the results. It seems reasonable in these patients to perform procedures to improve the clinical respiratory picture before intubation in less severe cases due to the aforementioned. Prone patient placement during invasive mechanical ventilation is a widespread practice in the management of severe ARDS of other etiologies. Currently, few attempts have been made to implement the prone position in patients who spontaneously ventilate with supplemental oxygen, high-flow nasal cannulas, or noninvasive mechanical ventilation. Taking into account that it is a procedure that does not require additional infrastructure within the services and does not represent an additional cost for its implementation, it becomes a valuable tool in the context of COVID-19 where intubation is associated with high mortality and in a Additionally, there are mechanical ventilator deficits in most hospitals. This work has feasibility to be carried out because it will be carried out in critical areas that have equipment and trained personnel for it in the different shifts, in addition to having patients diagnosed with COVID-19.

ELIGIBILITY:
Inclusion criteria

* Patient records with the following characteristics:
* Patients over 18 years of age
* Patients of both genders
* Patients diagnosed with COVID-19 infection
* Patients admitted to hospital
* Complete file

Non-inclusion criteria • Patients who do not decide to participate in the study

Exclusion criteria

• Files not found.

Elimination criteria

* Files with incomplete data
* File with a voluntary discharge or transfer note.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population Patients diagnosed with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 827 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
To analyze the relationship between the prone position and the need for orotracheal intubation. | 3 months
  Relationship between awake prone position and the tracheal intubation

SECONDARY OUTCOMES:
The impact of the prone position on the partial oxygen saturation / inspired oxygen fraction index (SaO2 / FiO2). | 3 months
  See the relationship between the awake prone position and the SaO2/FiO2 INDEX

OTHER OUTCOMES:
Determine the free hours without the need for orotracheal intubation of patients in the prone position. | 3 months
  Determine the free hours without the need for orotracheal intubation of patients in the prone position.

CONTACTS AND LOCATIONS:
Overall Officials: Orlando R Perez Nieto, MD, Principal Investigator — Hospital General San Juan del Rio
Locations (6):
- Mexico (6):
  - Hospital Materno Celaya, Celaya, Guanajuato
  - Hospital Santo Tomas, Querétaro City, Querétaro
  - Hospital General San Juan del Rio, Querétaro City, Querétaro
  - ISSSTE Hospital Regional Merida, Mérida, Yucatán
  - Hospital General de Zona 48 San PEDRO Xalpa IMSS, Estado de México
  - Hospital Fernando Quiroz Gutierrez, Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wan S, Li M, Ye Z, Yang C, Cai Q, Duan S, Song B. CT Manifestations and Clinical Characteristics of 1115 Patients with Coronavirus Disease 2019 (COVID-19): A Systematic Review and Meta-analysis. Acad Radiol. 2020 Jul;27(7):910-921. doi: 10.1016/j.acra.2020.04.033. Epub 2020 May 5. PMID 32505599
- [Result] Valter C, Christensen AM, Tollund C, Schonemann NK. Response to the prone position in spontaneously breathing patients with hypoxemic respiratory failure. Acta Anaesthesiol Scand. 2003 Apr;47(4):416-8. doi: 10.1034/j.1399-6576.2003.00088.x. PMID 12694139
- [Result] Scaravilli V, Grasselli G, Castagna L, Zanella A, Isgro S, Lucchini A, Patroniti N, Bellani G, Pesenti A. Prone positioning improves oxygenation in spontaneously breathing nonintubated patients with hypoxemic acute respiratory failure: A retrospective study. J Crit Care. 2015 Dec;30(6):1390-4. doi: 10.1016/j.jcrc.2015.07.008. Epub 2015 Jul 16. PMID 26271685
- [Result] Ding L, Wang L, Ma W, He H. Efficacy and safety of early prone positioning combined with HFNC or NIV in moderate to severe ARDS: a multi-center prospective cohort study. Crit Care. 2020 Jan 30;24(1):28. doi: 10.1186/s13054-020-2738-5. PMID 32000806
- [Result] Perez-Nieto OR, Guerrero-Gutierrez MA, Deloya-Tomas E, Namendys-Silva SA. Prone positioning combined with high-flow nasal cannula in severe noninfectious ARDS. Crit Care. 2020 Mar 23;24(1):114. doi: 10.1186/s13054-020-2821-y. No abstract available. PMID 32204726
- [Result] Sun Q, Qiu H, Huang M, Yang Y. Lower mortality of COVID-19 by early recognition and intervention: experience from Jiangsu Province. Ann Intensive Care. 2020 Mar 18;10(1):33. doi: 10.1186/s13613-020-00650-2. No abstract available. PMID 32189136
- [Result] Caputo ND, Strayer RJ, Levitan R. Early Self-Proning in Awake, Non-intubated Patients in the Emergency Department: A Single ED's Experience During the COVID-19 Pandemic. Acad Emerg Med. 2020 May;27(5):375-378. doi: 10.1111/acem.13994. PMID 32320506
- [Result] Slessarev M, Cheng J, Ondrejicka M, Arntfield R; Critical Care Western Research Group. Patient self-proning with high-flow nasal cannula improves oxygenation in COVID-19 pneumonia. Can J Anaesth. 2020 Sep;67(9):1288-1290. doi: 10.1007/s12630-020-01661-0. Epub 2020 Apr 21. No abstract available. PMID 32319029
- [Result] Lomoro P, Verde F, Zerboni F, Simonetti I, Borghi C, Fachinetti C, Natalizi A, Martegani A. COVID-19 pneumonia manifestations at the admission on chest ultrasound, radiographs, and CT: single-center study and comprehensive radiologic literature review. Eur J Radiol Open. 2020;7:100231. doi: 10.1016/j.ejro.2020.100231. Epub 2020 Apr 4. PMID 32289051
- [Result] Ai T, Yang Z, Hou H, Zhan C, Chen C, Lv W, Tao Q, Sun Z, Xia L. Correlation of Chest CT and RT-PCR Testing for Coronavirus Disease 2019 (COVID-19) in China: A Report of 1014 Cases. Radiology. 2020 Aug;296(2):E32-E40. doi: 10.1148/radiol.2020200642. Epub 2020 Feb 26. PMID 32101510
- [Derived] Perez-Nieto OR, Escarraman-Martinez D, Guerrero-Gutierrez MA, Zamarron-Lopez EI, Mancilla-Galindo J, Kammar-Garcia A, Martinez-Camacho MA, Deloya-Tomas E, Sanchez-Diaz JS, Macias-Garcia LA, Soriano-Orozco R, Cruz-Sanchez G, Salmeron-Gonzalez JD, Toledo-Rivera MA, Mata-Maqueda I, Morgado-Villasenor LA, Martinez-Mazariegos JJ, Flores Ramirez R, Medina-Estrada JL, Namendys-Silva SA; APRONOX Group. Awake prone positioning and oxygen therapy in patients with COVID-19: the APRONOX study. Eur Respir J. 2022 Feb 24;59(2):2100265. doi: 10.1183/13993003.00265-2021. Print 2022 Feb. PMID 34266942

DOCUMENTS (1):
  • Study Protocol (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT04407468/Prot_000.pdf